CLINICAL TRIAL: NCT05044325
Title: A Two-Part First Time in Human (FTIH) Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Repeat Oral Doses of GSK3884464 in a Randomized, Double Blind, Placebo-Controlled, Dose Escalation Study in Healthy Participants
Brief Title: A First Time in Human (FTIH) Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Repeat Doses of GSK3884464 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: To allow for additional assessments from supplementary non-clinical activities.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 213376
Record Dates: First submitted 2021-09-06; First posted 2021-09-14 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure
Keywords: First Time in Human; GSK3884464; Pharmacokinetics; Pharmacodynamics; Safety; Tolerability
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Part 1 Cohort 1 (C1): Placebo C1/ GSK3884464 3 milligrams (mg)/ GSK3884464 9mg (Experimental): Participants received GSK3884464 or placebo through oral administration in the treatment sequence: Placebo C1/ GSK3884464 3 milligrams (mg)/ GSK3884464 9mg across 3 treatment periods. There was a minimum of 7 days washout period between dosing in each session.
  Interventions: Drug: GSK3884464; Drug: Placebo
- Part 1 Cohort 1: GSK3884464 1 mg/ Placebo C1/ GSK3884464 9mg (Experimental): Participants received GSK3884464 or placebo through oral administration in the treatment sequence: GSK3884464 1 mg/ Placebo C1/ GSK3884464 9mg across 3 treatment periods. There was a minimum of 7 days washout period between dosing in each session.
  Interventions: Drug: GSK3884464; Drug: Placebo
- Part 1 Cohort 1: GSK3884464 1 mg/ GSK3884464 3 mg / Placebo C1 (Experimental): Participants received GSK3884464 or placebo through oral administration in the treatment sequence: GSK3884464 1 mg/ GSK3884464 3 mg / Placebo C1 across 3 treatment periods. There was a minimum of 7 days washout period between dosing in each session.
  Interventions: Drug: GSK3884464; Drug: Placebo
- Part 1 Cohort 2 (C2): Placebo C2/ GSK3884464 110 mg/ SD6 (Experimental): Participants received GSK3884464 or placebo through oral administration in the treatment sequence: Placebo C2/ GSK3884464 110 mg/ Single Dose (SD) 6 across 3 treatment periods. There was a minimum of 7 days washout period between dosing in each session.
  Interventions: Drug: GSK3884464; Drug: Placebo
- Part 1 Cohort 2: GSK3884464 30 mg/ Placebo C2/ SD6 (Experimental): Participants received GSK3884464 or placebo through oral administration in the treatment sequence: GSK3884464 30 mg/ Placebo C2/ SD6 across 3 treatment periods. There was a minimum of 7 days washout period between dosing in each session.
  Interventions: Drug: GSK3884464; Drug: Placebo
- Part 1 Cohort 2: GSK3884464 30 mg/ GSK3884464 110 mg / Placebo C2 (Experimental): Participants received GSK3884464 or placebo through oral administration in the treatment sequence: GSK3884464 30 mg/ GSK3884464 110 mg / Placebo C2 across 3 treatment periods. There was a minimum of 7 days washout period between dosing in each session.
  Interventions: Drug: GSK3884464; Drug: Placebo
- Part 1 Cohort 3 (C3): Placebo C3/ SD8/ SD9 (Experimental): Participants received GSK3884464 or placebo through oral administration in the treatment sequence: Placebo C3/ SD8/ SD9 across 3 treatment periods. There was a minimum of 7 days washout period between dosing in each session.
  Interventions: Drug: GSK3884464; Drug: Placebo
- Part 1 Cohort 3: GSK3884464 70 mg/ SD8/ Placebo C3 (Experimental): Participants received GSK3884464 or placebo through oral administration in the treatment sequence: GSK3884464 70 mg/ SD8/ Placebo C3 across 3 treatment periods. There was a minimum of 7 days washout period between dosing in each session.
  Interventions: Drug: GSK3884464; Drug: Placebo
- Part 2 Cohort 4 (C4): GSK3884464 15 mg (Experimental): Participants received GSK3884464 15 mg through oral administration.
  Interventions: Drug: GSK3884464
- Part 2 Cohort 4: Placebo C4 (Experimental): Participants received placebo through oral administration in Cohort 4.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3884464 — GSK3884464 will be administered
  Arms: Part 1 Cohort 1 (C1): Placebo C1/ GSK3884464 3 milligrams (mg)/ GSK3884464 9mg; Part 1 Cohort 1: GSK3884464 1 mg/ GSK3884464 3 mg / Placebo C1; Part 1 Cohort 1: GSK3884464 1 mg/ Placebo C1/ GSK3884464 9mg; Part 1 Cohort 2 (C2): Placebo C2/ GSK3884464 110 mg/ SD6; Part 1 Cohort 2: GSK3884464 30 mg/ GSK3884464 110 mg / Placebo C2; Part 1 Cohort 2: GSK3884464 30 mg/ Placebo C2/ SD6; Part 1 Cohort 3 (C3): Placebo C3/ SD8/ SD9; Part 1 Cohort 3: GSK3884464 70 mg/ SD8/ Placebo C3; Part 2 Cohort 4 (C4): GSK3884464 15 mg
Drug: Placebo — Placebo to match GSK3884464 will be administered.
  Arms: Part 1 Cohort 1 (C1): Placebo C1/ GSK3884464 3 milligrams (mg)/ GSK3884464 9mg; Part 1 Cohort 1: GSK3884464 1 mg/ GSK3884464 3 mg / Placebo C1; Part 1 Cohort 1: GSK3884464 1 mg/ Placebo C1/ GSK3884464 9mg; Part 1 Cohort 2 (C2): Placebo C2/ GSK3884464 110 mg/ SD6; Part 1 Cohort 2: GSK3884464 30 mg/ GSK3884464 110 mg / Placebo C2; Part 1 Cohort 2: GSK3884464 30 mg/ Placebo C2/ SD6; Part 1 Cohort 3 (C3): Placebo C3/ SD8/ SD9; Part 1 Cohort 3: GSK3884464 70 mg/ SD8/ Placebo C3; Part 2 Cohort 4: Placebo C4

SUMMARY:
This will be a FTIH study which aims to evaluate safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single and repeat oral doses of GSK3884464 administered to healthy participants.

ELIGIBILITY:
Inclusion criteria:

* Healthy as determined by the experienced investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring/assessment.
* Part 1: Body weight greater than or equal to (>=)50 kilograms (kg), body mass index (BMI) >=18 and less than or equal to (<=)30 kilograms per square meter (kg/m^2) (inclusive). Part 2: Body weight >=50 kg, BMI >=22 and <=30 kg/m^2 (inclusive).
* Participants with 18 to 50 years of age inclusive at the time of signing the informed consent.
* Male or females of non-childbearing potential.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion criteria:

* History or presence of significant cardiovascular, respiratory, hepatic, renal, gastrointestinal (Gastroesophageal reflux disease [GERD], nausea, vomiting or dysphagia), endocrine, hematological or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* History of current or past significant renal diseases.
* Clinically significant high blood pressure and/or history of hypertension as determined by the investigator.
* Serum troponin I or troponin-T greater than (>) the upper limit of normal (ULN).
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years.
* Any clinically relevant abnormality on the screening medical assessments.
* Alanine transaminase (ALT) > ULN.
* Bilirubin > ULN.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Unable to refrain from the use of prescription or non-prescription drug including vitamins, herbal and dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer [ for example (e.g.) Rifampin, St John's Wort extract]) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise participant safety. By exception, all participants may take Paracetamol (<=2 grams/day) up to 48 hours prior to the first dose of study drug.
* A positive laboratory confirmation of Coronavirus Disease-2019 (COVID-19) infection, or high clinical index of suspicion for COVID-19.
* Participants with Glycated hemoglobin (HbA1c) greater than (>)48 millimoles per mol (mmol/mol) at screening.
* Presence of Hepatitis B surface antigen at screening.
* Positive Hepatitis C antibody test result at screening.
* Positive Hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment.
* Positive pre-study drug/alcohol screen.
* Positive Human immunodeficiency virus (HIV) antibody test.
* Screening urine albumin to creatinine ratio >=30 milligrams/grams (mg/gm) (>=3 mg/mmol).
* Regular use of known drugs of abuse.
* Regular alcohol consumption within six months prior to the study defined as: An average weekly intake of >=14 units for males >=14 units for females. One unit is equivalent to 8 gm of alcohol: a half-pint (approximately 240 milliliters [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Smokelyzer test levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products (e.g.nicotine patches or vaporizing devices) within 3 months prior to screening.
* Participants with a history or current evidence of depression, bipolar disorder, suicidal ideation and behavior, or a lifetime history of suicide attempt will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 27 participants were enrolled in both Part 1 and Part 2 together.
Pre-assignment Details: This was a two parts study with single dose escalation in Part 1 and repeat dose in Part 2 in healthy participants. Part 1 was a 3-period crossover design with 3 cohorts, randomized to 3 periods in a 1:1:1 ratio. Within each period, allocation to GSK3884464 and placebo were a 2:1 ratio. Part 2 was a sequential design with 3 cohorts. The study was terminated after dosing 2 sentinel participants in Cohort 4 (which was first cohort to receive repeat doses). Hence, Cohort 5 and 6 were not conducted.
Period: Part A:Treatment Period 1
Arm/Group | Part 1 Cohort 1 (C1): Placebo C1/ GSK3884464 3 Milligrams (mg)/ GSK3884464 9mg | Part 1 Cohort 1: GSK3884464 1 mg/ Placebo C1/ GSK3884464 9mg | Part 1 Cohort 1: GSK3884464 1 mg/ GSK3884464 3 mg / Placebo C1 | Part 1 Cohort 2 (C2): Placebo C2/ GSK3884464 110 mg/ SD6 | Part 1 Cohort 2: GSK3884464 30 mg/ Placebo C2/ SD6 | Part 1 Cohort 2: GSK3884464 30 mg/ GSK3884464 110 mg / Placebo C2 | Part 1 Cohort 3 (C3): Placebo C3/ SD8/ SD9 | Part 1 Cohort 3: GSK3884464 70 mg/ SD8/ Placebo C3 | Part 2 Cohort 4 (C4): GSK3884464 15 mg | Part 2 Cohort 4: Placebo C4
Started | 3 | 3 | 3 | 3 | 3 | 3 | 1 | 1 | 0 | 0
Completed | 3 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 2 | 2 | 3 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Sponsor Terminated study treatment | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A:Treatment Period 2
Arm/Group | Part 1 Cohort 1 (C1): Placebo C1/ GSK3884464 3 Milligrams (mg)/ GSK3884464 9mg | Part 1 Cohort 1: GSK3884464 1 mg/ Placebo C1/ GSK3884464 9mg | Part 1 Cohort 1: GSK3884464 1 mg/ GSK3884464 3 mg / Placebo C1 | Part 1 Cohort 2 (C2): Placebo C2/ GSK3884464 110 mg/ SD6 | Part 1 Cohort 2: GSK3884464 30 mg/ Placebo C2/ SD6 | Part 1 Cohort 2: GSK3884464 30 mg/ GSK3884464 110 mg / Placebo C2 | Part 1 Cohort 3 (C3): Placebo C3/ SD8/ SD9 | Part 1 Cohort 3: GSK3884464 70 mg/ SD8/ Placebo C3 | Part 2 Cohort 4 (C4): GSK3884464 15 mg | Part 2 Cohort 4: Placebo C4
Started | 3 | 3 | 3 (New participant enrolled and dosed as a replacement of withdrawn participant.) | 1 | 2 | 2 | 0 | 0 | 0 | 0
Completed | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor Terminated study treatment | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part A:Treatment Period 3
Arm/Group | Part 1 Cohort 1 (C1): Placebo C1/ GSK3884464 3 Milligrams (mg)/ GSK3884464 9mg | Part 1 Cohort 1: GSK3884464 1 mg/ Placebo C1/ GSK3884464 9mg | Part 1 Cohort 1: GSK3884464 1 mg/ GSK3884464 3 mg / Placebo C1 | Part 1 Cohort 2 (C2): Placebo C2/ GSK3884464 110 mg/ SD6 | Part 1 Cohort 2: GSK3884464 30 mg/ Placebo C2/ SD6 | Part 1 Cohort 2: GSK3884464 30 mg/ GSK3884464 110 mg / Placebo C2 | Part 1 Cohort 3 (C3): Placebo C3/ SD8/ SD9 | Part 1 Cohort 3: GSK3884464 70 mg/ SD8/ Placebo C3 | Part 2 Cohort 4 (C4): GSK3884464 15 mg | Part 2 Cohort 4: Placebo C4
Started | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part 1 Cohort 1 (C1): Placebo C1/ GSK3884464 3 Milligrams (mg)/ GSK3884464 9mg | Part 1 Cohort 1: GSK3884464 1 mg/ Placebo C1/ GSK3884464 9mg | Part 1 Cohort 1: GSK3884464 1 mg/ GSK3884464 3 mg / Placebo C1 | Part 1 Cohort 2 (C2): Placebo C2/ GSK3884464 110 mg/ SD6 | Part 1 Cohort 2: GSK3884464 30 mg/ Placebo C2/ SD6 | Part 1 Cohort 2: GSK3884464 30 mg/ GSK3884464 110 mg / Placebo C2 | Part 1 Cohort 3 (C3): Placebo C3/ SD8/ SD9 | Part 1 Cohort 3: GSK3884464 70 mg/ SD8/ Placebo C3 | Part 2 Cohort 4 (C4): GSK3884464 15 mg | Part 2 Cohort 4: Placebo C4
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1 (C1): Placebo C1/ GSK3884464 3 Milligrams (mg)/ GSK3884464 9mg | Part 1 Cohort 1: GSK3884464 1 mg/ Placebo C1/ GSK3884464 9mg | Part 1 Cohort 1: GSK3884464 1 mg/ GSK3884464 3 mg / Placebo C1 | Part 1 Cohort 2 (C2): Placebo C2/ GSK3884464 110 mg/ SD6 | Part 1 Cohort 2: GSK3884464 30 mg/ Placebo C2/ SD6 | Part 1 Cohort 2: GSK3884464 30 mg/ GSK3884464 110 mg / Placebo C2 | Part 1 Cohort 3 (C3): Placebo C3/ SD8/ SD9 | Part 1 Cohort 3: GSK3884464 70 mg/ SD8/ Placebo C3 | Part 2 Cohort 4 (C4): GSK3884464 15 mg | Part 2 Cohort 4: Placebo C4 | Total
Number analyzed (Participants) | 3 | 4 | 4 | 3 | 4 | 5 | 1 | 1 | 1 | 1 | 27
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 30.3 (9.71) | 37.5 (6.61) | 36.5 (8.58) | 44.0 (6.08) | 31.8 (6.29) | 36.6 (6.15) | 37.0 | 36.0 | 24.0 | 46.0 | 36.0 (7.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 4 | 4 | 3 | 4 | 5 | 1 | 1 | 1 | 1 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3
  BLACK OR AFRICAN AMERICAN | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5
  WHITE | 3 | 1 | 2 | 2 | 3 | 4 | 1 | 0 | 0 | 1 | 17
  MULTIPLE | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Parts 1: Number of Participants With Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Time Frame: Up to Day 17
Population: The analysis was performed on the Safety Set that includes all randomized participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 Cohort 1: Placebo C1: Participants received placebo through oral administration in Cohort 1.
- Part 1 Cohort 1: GSK3884464 1 mg: Participants received GSK3884464 1 mg through oral administration.
- Part 1 Cohort 1: GSK3884464 3 mg: Participants received GSK3884464 3 mg through oral administration.
- Part 1 Cohort 1: GSK3884464 9 mg: Participants received GSK3884464 9 mg through oral administration.
- Part 1 Cohort 2: Placebo C2: Participants received placebo through oral administration in Cohort 2.
- Part 1 Cohort 2: GSK3884464 30 mg: Participants received GSK3884464 30 mg through oral administration.
- Part 1 Cohort 2: GSK3884464 110 mg: Participants received GSK3884464 110 mg through oral administration.
- Part 1 Cohort 3: Placebo C3: Participants received placebo through oral administration in Cohort 3.
- Part 1 Cohort 3: GSK3884464 70 mg: Participants received GSK3884464 70 mg through oral administration in Cohort 3.
Arm/Group | Part 1 Cohort 1: Placebo C1 | Part 1 Cohort 1: GSK3884464 1 mg | Part 1 Cohort 1: GSK3884464 3 mg | Part 1 Cohort 1: GSK3884464 9 mg | Part 1 Cohort 2: Placebo C2 | Part 1 Cohort 2: GSK3884464 30 mg | Part 1 Cohort 2: GSK3884464 110 mg | Part 1 Cohort 3: Placebo C3 | Part 1 Cohort 3: GSK3884464 70 mg
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5 | 6 | 3 | 1 | 1
Participants | 2 | 1 | 0 | 3 | 3 | 1 | 3 | 1 | 1

2. Primary Outcome: Parts 2: Number of Participants With Adverse Events (AEs)
Description: as for outcome 1
Time Frame: Up to Day 29
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Part 2 Cohort 4: GSK3884464 15 mg: Participants received GSK3884464 15 mg through oral administration in Cohort 4.
Arm/Group | Part 2 Cohort 4: Placebo C4 | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

3. Primary Outcome: Part 1: Number of Participants With Worst Case Chemistry Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected for analysis of chemistry parameters. PCI ranges were >2*Upper limit of normal (ULN) units per liter (U/L)(Alanine Aminotransferase [ALT]), >2*ULN (U/L) (Aspartate Aminotransferase ([AST]), >2*ULN (Alkaline Phosphatase [ALP]) (U/L), >1.5*ULN (micromoles per liter) (bilirubin), <2 or >2.75 millimoles/liter (L) (mmol/L)(calcium), <3 or >7.5 mmol/L (glucose), <3 or >5.3 mmol/L (potassium), <130 or >149 mmol/L (sodium). Participants were counted in worst case category that their value changes to (low, within [w/in] range or no change [NC], or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, are recorded in 'To within Range No Change' category. Participants were counted twice if participant had values that changed 'To Low' and 'To High', so percentages may not add to 100 percentage (%).
Time Frame: Up to Week 10
Population: The analysis was performed on the Safety Set that includes all randomized participants who received at least one dose of study intervention. Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: Placebo C1 | Part 1 Cohort 1: GSK3884464 1 mg | Part 1 Cohort 1: GSK3884464 3 mg | Part 1 Cohort 1: GSK3884464 9 mg | Part 1 Cohort 2: Placebo C2 | Part 1 Cohort 2: GSK3884464 30 mg | Part 1 Cohort 2: GSK3884464 110 mg | Part 1 Cohort 3: Placebo C3 | Part 1 Cohort 3: GSK3884464 70 mg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 5 | 6 | 3 | 1 | 1
Participants
  ALT, Period 1 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  ALT, Period 1 Worst Case Post-Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  ALT, Period 1 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  ALT, Period 1 Worst Case Post-Baseline, To W/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 0
  ALT, Period 1 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  ALT, Period 1 Worst Case Post-Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 1
  ALT, Period 2 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  ALT, Period 2 Worst Case Post-Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  ALT, Period 2 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  ALT, Period 2 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  | 6 |  | 2 |  | 1 |  |
  ALT, Period 2 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  ALT, Period 2 Worst Case Post-Baseline, To High | 0 |  | 0 |  | 0 |  | 2 |  |
  ALT, Period 3 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  ALT, Period 3 Worst Case Post-Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  ALT, Period 3 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  ALT, Period 3 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  ALT, Period 3 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  ALT, Period 3 Worst Case Post-Baseline, To High | 0 |  |  | 0 |  |  |  |  |
  AP, Period 1 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  AP, Period 1 Worst Case Post-Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  AP, Period 1 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  AP, Period 1 Worst Case Post-Baseline, To W/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 1
  AP, Period 1 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  AP, Period 1 Worst Case Post-Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  AP, Period 2 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  AP, Period 2 Worst Case Post-Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  AP, Period 2 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  AP, Period 2 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  AP, Period 2 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  AP, Period 2 Worst Case Post-Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  AP, Period 3 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  AP, Period 3 Worst Case Post-Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  AP, Period 3 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  AP, Period 3 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  AP, Period 3 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  AP, Period 3 Worst Case Post-Baseline, To High | 0 |  |  | 0 |  |  |  |  |
  AST, Period 1 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  AST, Period 1 Worst Case Post-Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  AST, Period 1 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  AST, Period 1 Worst Case Post-Baseline, To W/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 0
  AST, Period 1 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  AST, Period 1 Worst Case Post-Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 1
  AST, Period 2 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  AST, Period 2 Worst Case Post-Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  AST, Period 2 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  AST, Period 2 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  | 6 |  | 2 |  | 1 |  |
  AST, Period 2 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  AST, Period 2 Worst Case Post-Baseline, To High | 0 |  | 0 |  | 0 |  | 2 |  |
  AST, Period 3 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  AST, Period 3 Worst Case Post-Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  AST, Period 3 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  AST, Period 3 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  AST, Period 3 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  AST, Period 3 Worst Case Post-Baseline, To High | 0 |  |  | 0 |  |  |  |  |
  Bilirubin, Period 1 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Bilirubin, Period 1 Worst Case Post-Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Bilirubin, Period 1 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Bilirubin, Period 1 Worst Case Post-Baseline, To W/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 1
  Bilirubin, Period 1 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Bilirubin, Period 1 Worst Case Post-Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Bilirubin, Period 2 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Bilirubin, Period 2 Worst Case Post-Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  Bilirubin, Period 2 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Bilirubin, Period 2 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  Bilirubin, Period 2 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Bilirubin, Period 2 Worst Case Post-Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  Bilirubin, Period 3 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Bilirubin, Period 3 Worst Case Post-Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  Bilirubin, Period 3 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Bilirubin, Period 3 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  Bilirubin, Period 3 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Bilirubin, Period 3 Worst Case Post-Baseline, To High | 0 |  |  | 0 |  |  |  |  |
  Calcium, Period 1 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Calcium, Period 1 Worst Case Post-Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Calcium, Period 1 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Calcium, Period 1 Worst Case Post-Baseline, To W/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 1
  Calcium, Period 1 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Calcium, Period 1 Worst Case Post-Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Calcium, Period 2 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Calcium, Period 2 Worst Case Post-Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  Calcium, Period 2 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Calcium, Period 2 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  Calcium, Period 2 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Calcium, Period 2 Worst Case Post-Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  Calcium, Period 3 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Calcium, Period 3 Worst Case Post-Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  Calcium, Period 3 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Calcium, Period 3 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  Calcium, Period 3 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Calcium, Period 3 Worst Case Post-Baseline, To High | 0 |  |  | 0 |  |  |  |  |
  Glucose, Period 1 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Glucose, Period 1 Worst Case Post-Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Glucose, Period 1 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Glucose, Period 1 Worst Case Post-Baseline, To W/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 1
  Glucose, Period 1 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Glucose, Period 1 Worst Case Post-Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Glucose, Period 2 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Glucose, Period 2 Worst Case Post-Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  Glucose, Period 2 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Glucose, Period 2 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  Glucose, Period 2 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Glucose, Period 2 Worst Case Post-Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  Glucose, Period 3 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Glucose, Period 3 Worst Case Post-Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  Glucose, Period 3 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Glucose, Period 3 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  Glucose, Period 3 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Glucose, Period 3 Worst Case Post-Baseline, To High | 0 |  |  | 0 |  |  |  |  |
  Potassium, Period 1 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Potassium, Period 1 Worst Case Post-Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Potassium, Period 1 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Potassium, Period 1 Worst Case Post-Baseline, To W/in Range or No Change | 3 | 6 |  |  | 3 | 5 |  | 1 | 1
  Potassium, Period 1 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Potassium, Period 1 Worst Case Post-Baseline, To High | 0 | 0 |  |  | 0 | 1 |  | 0 | 0
  Potassium, Period 2 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Potassium, Period 2 Worst Case Post-Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  Potassium, Period 2 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Potassium, Period 2 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  Potassium, Period 2 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Potassium, Period 2 Worst Case Post-Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  Potassium, Period 3 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Potassium, Period 3 Worst Case Post-Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  Potassium, Period 3 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Potassium, Period 3 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  |  | 5 |  |  |  |  |
  Potassium, Period 3 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Potassium, Period 3 Worst Case Post-Baseline, To High | 0 |  |  | 1 |  |  |  |  |
  Sodium, Period 1 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Sodium, Period 1 Worst Case Post-Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Sodium, Period 1 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Sodium, Period 1 Worst Case Post-Baseline, To W/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 1
  Sodium, Period 1 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Sodium, Period 1 Worst Case Post-Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Sodium, Period 2 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Sodium, Period 2 Worst Case Post-Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  Sodium, Period 2 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Sodium, Period 2 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  Sodium, Period 2 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Sodium, Period 2 Worst Case Post-Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  Sodium, Period 3 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Sodium, Period 3 Worst Case Post-Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  Sodium, Period 3 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Sodium, Period 3 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  Sodium, Period 3 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Sodium, Period 3 Worst Case Post-Baseline, To High | 0 |  |  | 0 |  |  |  |  |

4. Primary Outcome: Part 1: Number of Participants With Worst Case Hematology Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected for analysis of hematology parameters. The ranges for hematology parameters are as follows: Hematocrit[>51 percent(%)-male, >45%-female], Hemoglobin [Higher: >175 grams/Liter(g/L) in male, >150g/L in female and Low: less than(<) 100g/L in male, <95g/L in female], Lymphocytes[<0.97 10^9/L], Neutrophils[<1.5 10^9/L], Platelets[High: >550 10^9/ L and Low: <100 10^9/ L], White blood cells[High:>18 10^9/L Low:<2 10^9/L], Red blood cells[Low: <3.0 10^12/L in male, <2.5 10^12/L]. Participants were counted in worst case category that their value changes to (low, within range [W/in] or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (for example-High to High), or whose value became within range, were recorded in "To within Range or No Change" category. Participants were counted twice if participant has values that changed 'To Low' & 'To High', so the percentages may not add to 100%.
Time Frame: Up to Week 10
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: Placebo C1 | Part 1 Cohort 1: GSK3884464 1 mg | Part 1 Cohort 1: GSK3884464 3 mg | Part 1 Cohort 1: GSK3884464 9 mg | Part 1 Cohort 2: Placebo C2 | Part 1 Cohort 2: GSK3884464 30 mg | Part 1 Cohort 2: GSK3884464 110 mg | Part 1 Cohort 3: Placebo C3 | Part 1 Cohort 3: GSK3884464 70 mg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 5 | 6 | 3 | 1 | 1
Participants
  Erythrocytes, Period 1 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Erythrocytes, Period 1 Worst Case Post-Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Erythrocytes, Period 1 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Erythrocytes, Period 1 Worst Case Post-Baseline, To W/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 1
  Erythrocytes, Period 1 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Erythrocytes, Period 1 Worst Case Post-Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Erythrocytes, Period 2 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Erythrocytes, Period 2 Worst Case Post-Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  Erythrocytes, Period 2 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Erythrocytes, Period 2 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  Erythrocytes, Period 2 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Erythrocytes, Period 2 Worst Case Post-Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  Erythrocytes, Period 3 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Erythrocytes, Period 3 Worst Case Post-Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  Erythrocytes, Period 3 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Erythrocytes, Period 3 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  Erythrocytes, Period 3 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Erythrocytes, Period 3 Worst Case Post-Baseline, To High | 0 |  |  | 0 |  |  |  |  |
  Hematocrit, Period 1 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Hematocrit, Period 1 Worst Case Post-Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Hematocrit, Period 1 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Hematocrit, Period 1 Worst Case Post-Baseline, To W/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 1
  Hematocrit, Period 1 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Hematocrit, Period 1 Worst Case Post-Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Hematocrit, Period 2 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Hematocrit, Period 2 Worst Case Post-Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  Hematocrit, Period 2 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Hematocrit, Period 2 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  Hematocrit, Period 2 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Hematocrit, Period 2 Worst Case Post-Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  Hematocrit, Period 3 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Hematocrit, Period 3 Worst Case Post-Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  Hematocrit, Period 3 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Hematocrit, Period 3 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  Hematocrit, Period 3 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Hematocrit, Period 3 Worst Case Post-Baseline, To High | 0 |  |  | 0 |  |  |  |  |
  Hemoglobin, Period 1 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Hemoglobin, Period 1 Worst Case Post-Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Hemoglobin, Period 1 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Hemoglobin, Period 1 Worst Case Post-Baseline, To W/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 1
  Hemoglobin, Period 1 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Hemoglobin, Period 1 Worst Case Post-Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Hemoglobin, Period 2 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Hemoglobin, Period 2 Worst Case Post-Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  Hemoglobin, Period 2 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Hemoglobin, Period 2 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  Hemoglobin, Period 2 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Hemoglobin, Period 2 Worst Case Post-Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  Hemoglobin, Period 3 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, Period 3 Worst Case Post-Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  Hemoglobin, Period 3 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, Period 3 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  Hemoglobin, Period 3 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, Period 3 Worst Case Post-Baseline, To High | 0 |  |  | 0 |  |  |  |  |
  Leukocytes, Period 1 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Leukocytes, Period 1 Worst Case Post-Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Leukocytes, Period 1 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Leukocytes, Period 1 Worst Case Post-Baseline, To W/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 1
  Leukocytes, Period 1 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Leukocytes, Period 1 Worst Case Post-Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Leukocytes, Period 2 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Leukocytes, Period 2 Worst Case Post-Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  Leukocytes, Period 2 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Leukocytes, Period 2 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  Leukocytes, Period 2 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Leukocytes, Period 2 Worst Case Post-Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  Leukocytes, Period 3 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Leukocytes, Period 3 Worst Case Post-Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  Leukocytes, Period 3 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Leukocytes, Period 3 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  Leukocytes, Period 3 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Leukocytes, Period 3 Worst Case Post-Baseline, To High | 0 |  |  | 0 |  |  |  |  |
  Neutrophils, Period 1 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Neutrophils, Period 1 Worst Case Post-Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Neutrophils, Period 1 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Neutrophils, Period 1 Worst Case Post-Baseline, To W/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 1
  Neutrophils, Period 1 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Neutrophils, Period 1 Worst Case Post-Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Neutrophils, Period 2 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Neutrophils, Period 2 Worst Case Post-Baseline, To Low | 0 |  | 0 |  | 1 |  | 0 |  |
  Neutrophils, Period 2 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Neutrophils, Period 2 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  | 6 |  | 1 |  | 3 |  |
  Neutrophils, Period 2 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Neutrophils, Period 2 Worst Case Post-Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  Neutrophils, Period 3 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Neutrophils, Period 3 Worst Case Post-Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  Neutrophils, Period 3 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Neutrophils, Period 3 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  Neutrophils, Period 3 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Neutrophils, Period 3 Worst Case Post-Baseline, To High | 0 |  |  | 0 |  |  |  |  |
  Platelets, Period 1 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Platelets, Period 1 Worst Case Post-Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Platelets, Period 1 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Platelets, Period 1 Worst Case Post-Baseline, To W/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 1
  Platelets, Period 1 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Platelets, Period 1 Worst Case Post-Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Platelets, Period 2 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Platelets, Period 2 Worst Case Post-Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  Platelets, Period 2 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Platelets, Period 2 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  Platelets, Period 2 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Platelets, Period 2 Worst Case Post-Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  Platelets, Period 3 Worst Case Post-Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Platelets, Period 3 Worst Case Post-Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  Platelets, Period 3 Worst Case Post-Baseline, To W/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Platelets, Period 3 Worst Case Post-Baseline, To W/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  Platelets, Period 3 Worst Case Post-Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Platelets, Period 3 Worst Case Post-Baseline, To High | 0 |  |  | 0 |  |  |  |  |

5. Primary Outcome: Part 1: Number of Participants With Worst Case Urinalysis Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: Urine samples were collected to assess urine glucose, protein and ketones using dipstick method. The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters were recorded as negative, trace, 1+, 2+, 3+ indicating proportional concentrations in the urine sample. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Result for urinalysis parameters were recorded as no change/decreased and any increase.
Time Frame: Up to Week 10
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: Placebo C1 | Part 1 Cohort 1: GSK3884464 1 mg | Part 1 Cohort 1: GSK3884464 3 mg | Part 1 Cohort 1: GSK3884464 9 mg | Part 1 Cohort 2: Placebo C2 | Part 1 Cohort 2: GSK3884464 30 mg | Part 1 Cohort 2: GSK3884464 110 mg | Part 1 Cohort 3: Placebo C3 | Part 1 Cohort 3: GSK3884464 70 mg
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5 | 6 | 3 | 1 | 1
Participants
  Glucose, No Change/Decreased | 9 | 6 | 6 | 6 | 5 | 6 | 3 | 1 | 1
  Ketones, No Change/Decreased | 9 | 6 | 6 | 6 | 5 | 6 | 3 | 1 | 1
  Protein, No Change/Decreased | 9 | 6 | 6 | 6 | 5 | 5 | 3 | 1 | 1
  Protein, Increase to TRACE | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

6. Primary Outcome: Part 1: Number of Participants With Clinically Significant Changes in Hepatobiliary Laboratory Values
Description: Blood samples were collected to evaluate hepatobiliary abnormalities. Number of participants with Bilirubin (BIL), Alkaline phosphatase (ALP), Alanine Aminotransferase (ALT)/combination of these with levels more than the defined hepatobiliary abnormality criteria were presented. Hepatocellular injury is defined as ([ALT/ALT ULN]/[ALP/ALP ULN]) >= 5 and ALT >=3xULN.
Time Frame: Up to Week 10
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: Placebo C1 | Part 1 Cohort 1: GSK3884464 1 mg | Part 1 Cohort 1: GSK3884464 3 mg | Part 1 Cohort 1: GSK3884464 9 mg | Part 1 Cohort 2: Placebo C2 | Part 1 Cohort 2: GSK3884464 30 mg | Part 1 Cohort 2: GSK3884464 110 mg | Part 1 Cohort 3: Placebo C3 | Part 1 Cohort 3: GSK3884464 70 mg
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5 | 6 | 3 | 1 | 1
Participants
  ALT >=3xULN and BIL >=2xULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT >3xULN and BIL >= 2xULN and (ALP <2xULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT >3xULN and INR >1.5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
  ALT >3xULN and INR >1.5 |  |  |  |  |  |  | 0 |  |
  Hepatocellular injury | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hepatocellular injury and BIL >2xULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT > 1.5xULN | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
  ALT >= 3xULN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  ALT >= 5xULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT >= 8xULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT >= 10xULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT >= 20xULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Part 1: Number of Participants With Clinically Significant Changes in 12-lead Electrocardiogram (ECG) Laboratory Values
Description: Twelve lead ECG was obtained using an ECG machine that automatically calculated the heart rate and measured QTc, PR, QRS intervals. Abnormal findings were categorized as clinically significant and not clinically significant. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for number of participants with worst case post-Baseline abnormal ECG findings have been presented.
Time Frame: Up to Week 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: Placebo C1 | Part 1 Cohort 1: GSK3884464 1 mg | Part 1 Cohort 1: GSK3884464 3 mg | Part 1 Cohort 1: GSK3884464 9 mg | Part 1 Cohort 2: Placebo C2 | Part 1 Cohort 2: GSK3884464 30 mg | Part 1 Cohort 2: GSK3884464 110 mg | Part 1 Cohort 3: Placebo C3 | Part 1 Cohort 3: GSK3884464 70 mg
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5 | 6 | 3 | 1 | 1
Participants
  Period 1 Day -1, Not Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day -1, Not Clinically Significant | 1 | 5 |  |  | 0 | 2 |  | 0 | 0
  Period 1 Day -1, Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day -1, Clinically Significant | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Period 1 Day 1, Not Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day 1, Not Clinically Significant | 1 | 3 |  |  | 1 | 1 |  | 0 | 0
  Period 1 Day 1, Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day 1, Clinically Significant | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Period 1 Day 2, Not Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day 2, Not Clinically Significant | 0 | 0 |  |  | 0 | 1 |  | 0 | 0
  Period 1 Day 2, Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day 2, Clinically Significant | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Period 1 Day 3, Not Clinically Significant: number analyzed (Participants) | 3 | 5 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day 3, Not Clinically Significant | 0 | 0 |  |  | 0 | 1 |  | 0 | 0
  Period 1 Day 3, Clinically Significant: number analyzed (Participants) | 3 | 5 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day 3, Clinically Significant | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Period 1 Day 4, Not Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day 4, Not Clinically Significant | 0 | 0 |  |  | 1 | 2 |  | 0 | 0
  Period 1 Day 4, Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day 4, Clinically Significant | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Period 1 Day 5, Not Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day 5, Not Clinically Significant | 0 | 1 |  |  | 0 | 2 |  | 0 | 0
  Period 1 Day 5, Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day 5, Clinically Significant | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Period 1 Day 6, Not Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day 6, Not Clinically Significant | 0 | 1 |  |  | 1 | 2 |  | 0 | 0
  Period 1 Day 6, Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day 6, Clinically Significant | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Period 2 Day -1, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day -1, Not Clinically Significant | 1 |  | 1 |  | 2 |  | 0 |  |
  Period 2 Day -1, Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day -1, Clinically Significant | 0 |  | 0 |  | 0 |  | 0 |  |
  Period 2 Day 1, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 1, Not Clinically Significant | 0 |  | 2 |  | 1 |  | 0 |  |
  Period 2 Day 1, Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 1, Clinically Significant | 0 |  | 0 |  | 0 |  | 0 |  |
  Period 2 Day 2, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 2, Not Clinically Significant | 0 |  | 1 |  | 0 |  | 0 |  |
  Period 2 Day 2, Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 2, Clinically Significant | 0 |  | 0 |  | 0 |  | 0 |  |
  Period 2 Day 3, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 3, Not Clinically Significant | 1 |  | 2 |  | 2 |  | 0 |  |
  Period 2 Day 3, Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 3, Clinically Significant | 0 |  | 0 |  | 0 |  | 0 |  |
  Period 2 Day 4, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 4, Not Clinically Significant | 1 |  | 0 |  | 0 |  | 0 |  |
  Period 2 Day 4, Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 4, Clinically Significant | 0 |  | 0 |  | 0 |  | 0 |  |
  Period 2 Day 5, Not Clinically Significant: number analyzed (Participants) | 2 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 5, Not Clinically Significant | 0 |  | 0 |  | 1 |  | 0 |  |
  Period 2 Day 5, Clinically Significant: number analyzed (Participants) | 2 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 5, Clinically Significant | 0 |  | 0 |  | 0 |  | 0 |  |
  Period 2 Day 6, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 6, Not Clinically Significant | 3 |  | 2 |  | 0 |  | 0 |  |
  Period 2 Day 6, Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 6, Clinically Significant | 0 |  | 0 |  | 0 |  | 0 |  |
  Period 3 Day -1, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day -1, Not Clinically Significant | 2 |  |  | 1 |  |  |  |  |
  Period 3 Day -1, Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day -1, Clinically Significant | 0 |  |  | 0 |  |  |  |  |
  Period 3 Day 1, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 1, Not Clinically Significant | 3 |  |  | 6 |  |  |  |  |
  Period 3 Day 1, Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 1, Clinically Significant | 0 |  |  | 0 |  |  |  |  |
  Period 3 Day 2, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 2, Not Clinically Significant | 0 |  |  | 1 |  |  |  |  |
  Period 3 Day 2, Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 2, Clinically Significant | 0 |  |  | 0 |  |  |  |  |
  Period 3 Day 3, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 3, Not Clinically Significant | 1 |  |  | 0 |  |  |  |  |
  Period 3 Day 3, Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 3, Clinically Significant | 0 |  |  | 0 |  |  |  |  |
  Period 3 Day 4, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 4, Not Clinically Significant | 1 |  |  | 1 |  |  |  |  |
  Period 3 Day 4, Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 4, Clinically Significant | 0 |  |  | 0 |  |  |  |  |
  Period 3 Day 5, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 5, Not Clinically Significant | 1 |  |  | 2 |  |  |  |  |
  Period 3 Day 5, Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 5, Clinically Significant | 0 |  |  | 0 |  |  |  |  |
  Period 3 Day 6, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 6, Not Clinically Significant | 0 |  |  | 1 |  |  |  |  |
  Period 3 Day 6, Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 6, Clinically Significant | 0 |  |  | 0 |  |  |  |  |
  Worst Case Post Baseline, Not Clinically Significant | 8 | 6 | 5 | 6 | 4 | 5 | 0 | 0 | 0
  Worst Case Post Baseline, Clinically Significant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Part 1: Number of Participants With Worst Case Vital Signs Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: Vital signs included diastolic blood pressure (DBP), systolic blood pressure (SBP), pulse rate (PR), body temperature, respiratory rate (RR) and were measured after resting for at least 5 minutes in semi-supine position. PCI ranges were, SBP (millimeters of mercury[mmHg]): <85 (low) or >160 (high), DBP (mmHg): <45 (low) or >100 (high), heart rate (beats per minute): <40 (low) or >110 (high), respiration rate (breaths per minute):<=8 (low) or >20 (high) and body temperature (degrees Celsius) <=35.5 (low) or >38.0 (high). Participants were counted in worst case category that their value changes to (low, within range or no change, or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, are recorded in 'To W/in Range No Change' category. Participants were counted twice if participant had values that changed 'To Low' and 'To High', so percentages may not add to 100%.
Time Frame: Up to Week 10
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: Placebo C1 | Part 1 Cohort 1: GSK3884464 1 mg | Part 1 Cohort 1: GSK3884464 3 mg | Part 1 Cohort 1: GSK3884464 9 mg | Part 1 Cohort 2: Placebo C2 | Part 1 Cohort 2: GSK3884464 30 mg | Part 1 Cohort 2: GSK3884464 110 mg | Part 1 Cohort 3: Placebo C3 | Part 1 Cohort 3: GSK3884464 70 mg
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5 | 6 | 3 | 1 | 1
Participants
  DBP, Period 1 Worst Case Post Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  DBP, Period 1 Worst Case Post Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  DBP, Period 1 Worst Case Post Baseline, To w/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  DBP, Period 1 Worst Case Post Baseline, To w/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 1
  DBP, Period 1 Worst Case Post Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  DBP, Period 1 Worst Case Post Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  DBP, Period 2 Worst Case Post Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  DBP, Period 2 Worst Case Post Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  DBP, Period 2 Worst Case Post Baseline, To w/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  DBP, Period 2 Worst Case Post Baseline, To w/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  DBP, Period 2 Worst Case Post Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  DBP, Period 2 Worst Case Post Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  DBP, Period 3 Worst Case Post Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  DBP, Period 3 Worst Case Post Baseline, To Low | 1 |  |  | 0 |  |  |  |  |
  DBP, Period 3 Worst Case Post Baseline, To w/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  DBP, Period 3 Worst Case Post Baseline, To w/in Range or No Change | 2 |  |  | 6 |  |  |  |  |
  DBP, Period 3 Worst Case Post Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  DBP, Period 3 Worst Case Post Baseline, To High | 0 |  |  | 0 |  |  |  |  |
  PR, Period 1 Worst Case Post Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  PR, Period 1 Worst Case Post Baseline, To Low | 1 | 1 |  |  | 0 | 1 |  | 0 | 0
  PR, Period 1 Worst Case Post Baseline, To w/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  PR, Period 1 Worst Case Post Baseline, To w/in Range or No Change | 2 | 5 |  |  | 3 | 5 |  | 1 | 1
  PR, Period 1 Worst Case Post Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  PR, Period 1 Worst Case Post Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  PR, Period 2 Worst Case Post Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  PR, Period 2 Worst Case Post Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  PR, Period 2 Worst Case Post Baseline, To w/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  PR, Period 2 Worst Case Post Baseline, To w/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  PR, Period 2 Worst Case Post Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  PR, Period 2 Worst Case Post Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  PR, Period 3 Worst Case Post Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  PR, Period 3 Worst Case Post Baseline, To Low | 0 |  |  | 1 |  |  |  |  |
  PR, Period 3 Worst Case Post Baseline, To w/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  PR, Period 3 Worst Case Post Baseline, To w/in Range or No Change | 3 |  |  | 5 |  |  |  |  |
  PR, Period 3 Worst Case Post Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  PR, Period 3 Worst Case Post Baseline, To High | 0 |  |  | 0 |  |  |  |  |
  Systolic Blood Pressure, Period 1 Worst Case Post Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Systolic Blood Pressure, Period 1 Worst Case Post Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Systolic Blood Pressure, Period 1 Worst Case Post Baseline, To w/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Systolic Blood Pressure, Period 1 Worst Case Post Baseline, To w/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 1
  Systolic Blood Pressure, Period 1 Worst Case Post Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Systolic Blood Pressure, Period 1 Worst Case Post Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Systolic Blood Pressure, Period 2 Worst Case Post Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Systolic Blood Pressure, Period 2 Worst Case Post Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  Systolic Blood Pressure, Period 2 Worst Case Post Baseline, To w/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Systolic Blood Pressure, Period 2 Worst Case Post Baseline, To w/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  Systolic Blood Pressure, Period 2 Worst Case Post Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Systolic Blood Pressure, Period 2 Worst Case Post Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  Systolic Blood Pressure, Period 3 Worst Case Post Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure, Period 3 Worst Case Post Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  Systolic Blood Pressure, Period 3 Worst Case Post Baseline, To w/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure, Period 3 Worst Case Post Baseline, To w/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  Systolic Blood Pressure, Period 3 Worst Case Post Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure, Period 3 Worst Case Post Baseline, To High | 0 |  |  | 0 |  |  |  |  |
  RR, Period 1 Worst Case Post Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  RR, Period 1 Worst Case Post Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  RR, Period 1 Worst Case Post Baseline, To w/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  RR, Period 1 Worst Case Post Baseline, To w/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 1
  RR, Period 1 Worst Case Post Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  RR, Period 1 Worst Case Post Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  RR, Period 2 Worst Case Post Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  RR, Period 2 Worst Case Post Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  RR, Period 2 Worst Case Post Baseline, To w/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  RR, Period 2 Worst Case Post Baseline, To w/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  RR, Period 2 Worst Case Post Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  RR, Period 2 Worst Case Post Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  RR, Period 3 Worst Case Post Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  RR, Period 3 Worst Case Post Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  RR, Period 3 Worst Case Post Baseline, To w/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  RR, Period 3 Worst Case Post Baseline, To w/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  RR, Period 3 Worst Case Post Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  RR, Period 3 Worst Case Post Baseline, To High | 0 |  |  | 0 |  |  |  |  |
  Temperature, Period 1 Worst Case Post Baseline, To Low: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Temperature, Period 1 Worst Case Post Baseline, To Low | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Temperature, Period 1 Worst Case Post Baseline, To w/in Range or No Change: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Temperature, Period 1 Worst Case Post Baseline, To w/in Range or No Change | 3 | 6 |  |  | 3 | 6 |  | 1 | 1
  Temperature, Period 1 Worst Case Post Baseline, To High: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Temperature, Period 1 Worst Case Post Baseline, To High | 0 | 0 |  |  | 0 | 0 |  | 0 | 0
  Temperature, Period 2 Worst Case Post Baseline, To Low: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Temperature, Period 2 Worst Case Post Baseline, To Low | 0 |  | 0 |  | 0 |  | 0 |  |
  Temperature, Period 2 Worst Case Post Baseline, To w/in Range or No Change: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Temperature, Period 2 Worst Case Post Baseline, To w/in Range or No Change | 3 |  | 6 |  | 2 |  | 3 |  |
  Temperature, Period 2 Worst Case Post Baseline, To High: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Temperature, Period 2 Worst Case Post Baseline, To High | 0 |  | 0 |  | 0 |  | 0 |  |
  Temperature, Period 3 Worst Case Post Baseline, To Low: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Temperature, Period 3 Worst Case Post Baseline, To Low | 0 |  |  | 0 |  |  |  |  |
  Temperature, Period 3 Worst Case Post Baseline, To w/in Range or No Change: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Temperature, Period 3 Worst Case Post Baseline, To w/in Range or No Change | 3 |  |  | 6 |  |  |  |  |
  Temperature, Period 3 Worst Case Post Baseline, To High: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Temperature, Period 3 Worst Case Post Baseline, To High | 0 |  |  | 0 |  |  |  |  |

9. Primary Outcome: Part 1: Number of Participants With Clinically Significant Changes in Continuous Telemetry
Description: Continuous cardiac telemetry was performed in a supine position after at least 5 minutes of rest. Number of participants who had abnormal findings upon cardiac telemetry assessment have been presented.
Time Frame: Upto Day 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: Placebo C1 | Part 1 Cohort 1: GSK3884464 1 mg | Part 1 Cohort 1: GSK3884464 3 mg | Part 1 Cohort 1: GSK3884464 9 mg | Part 1 Cohort 2: Placebo C2 | Part 1 Cohort 2: GSK3884464 30 mg | Part 1 Cohort 2: GSK3884464 110 mg | Part 1 Cohort 3: Placebo C3 | Part 1 Cohort 3: GSK3884464 70 mg
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5 | 6 | 3 | 1 | 1
Participants
  Period 1 Day 2, Not Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 0
  Period 1 Day 2, Not Clinically Significant | 1 | 0 |  |  | 0 | 0 |  | 0 |
  Period 1 Day 2, Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 0
  Period 1 Day 2, Clinically Significant | 0 | 0 |  |  | 0 | 1 |  | 0 |
  Period 1 Day 3, Not Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day 3, Not Clinically Significant | 1 | 0 |  |  | 0 | 0 |  | 0 | 1
  Period 1 Day 3, Clinically Significant: number analyzed (Participants) | 3 | 6 | 0 | 0 | 3 | 6 | 0 | 1 | 1
  Period 1 Day 3, Clinically Significant | 0 | 0 |  |  | 0 | 1 |  | 0 | 0
  Period 2 Day 2, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 2, Not Clinically Significant | 2 |  | 3 |  | 1 |  | 1 |  |
  Period 2 Day 2, Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 2, Clinically Significant | 0 |  | 0 |  | 0 |  | 0 |  |
  Period 2 Day 3, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 3, Not Clinically Significant | 2 |  | 3 |  | 1 |  | 1 |  |
  Period 2 Day 3, Clinically Significant: number analyzed (Participants) | 3 | 0 | 6 | 0 | 2 | 0 | 3 | 0 | 0
  Period 2 Day 3, Clinically Significant | 0 |  | 0 |  | 0 |  | 0 |  |
  Period 3 Day 2, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 2, Not Clinically Significant | 1 |  |  | 1 |  |  |  |  |
  Period 3 Day 2, Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 2, Clinically Significant | 0 |  |  | 0 |  |  |  |  |
  Period 3 Day 3, Not Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 3, Not Clinically Significant | 1 |  |  | 1 |  |  |  |  |
  Period 3 Day 3, Clinically Significant: number analyzed (Participants) | 3 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  Period 3 Day 3, Clinically Significant | 0 |  |  | 0 |  |  |  |  |
  Worst Case Post Baseline, Not Clinically Significant | 4 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 1
  Worst Case Post Baseline, Clinically Significant | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

10. Primary Outcome: Part 2: Cohorts 4: Number of Participants With Worst Case Chemistry Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected for analysis of chemistry parameters. PCI ranges were >=2*Upper limit of normal (ULN) units per liter (U/L)(Alanine Aminotransferase [ALT]), >=2*ULN (U/L) (Aspartate Aminotransferase ([AST]), >=2*ULN (Alkaline Phosphatase [ALP]) (U/L), >=1.5*ULN (micromoles per liter) (bilirubin), <2 or >2.75 millimoles/liter (L) (mmol/L)(calcium), <3 or >11 mmol/L (glucose), <3 or >5.5 mmol/L (potassium), <130 or >150 mmol/L (sodium),<50 or >85 grams/liter (protein). Participants were counted in worst case category that their value changes to (low, within [w/in] range or no change [NC], or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, are recorded in 'To within Range No Change' category. Participants were counted twice if participant had values that changed 'To Low' and 'To High', so percentages may not add to 100 percentage (%)
Time Frame: Upto Week 9
Population: The analysis was performed on the Safety Set that includes all randomized participants who received at least one dose of study intervention. The study was terminated after dosing 2 sentinel participants in Cohort 4. Hence Cohort 5 and 6 were not conducted.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 4: Placebo C4 | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1 | 1
Participants
  ALT, Worst Case Post-Baseline, To Low | 0 | 0
  ALT, Worst Case Post-Baseline, To W/in Range or No Change | 1 | 0
  ALT, Worst Case Post-Baseline, To High | 0 | 1
  AP, Worst Case Post-Baseline, To Low | 0 | 0
  AP, Worst Case Post-Baseline, To W/in Range or No Change | 1 | 1
  AP, Worst Case Post-Baseline, To High | 0 | 0
  AST, Worst Case Post-Baseline, To Low | 0 | 0
  AST, Worst Case Post-Baseline, To W/in Range or No Change | 1 | 1
  AST, Worst Case Post-Baseline, To High | 0 | 0
  Bilirubin, Worst Case Post-Baseline, To Low | 0 | 0
  Bilirubin, Worst Case Post-Baseline, To W/in Range or No Change | 1 | 1
  Bilirubin, Worst Case Post-Baseline, To High | 0 | 0
  Calcium, Worst Case Post-Baseline, To Low | 0 | 0
  Calcium, Worst Case Post-Baseline, To W/in Range or No Change | 1 | 1
  Calcium, Worst Case Post-Baseline, To High | 0 | 0
  Glucose, Worst Case Post-Baseline, To Low | 0 | 0
  Glucose, Worst Case Post-Baseline, To W/in Range or No Change | 1 | 1
  Glucose, Worst Case Post-Baseline, To High | 0 | 0
  Potassium, Worst Case Post-Baseline, To Low | 0 | 0
  Potassium, Worst Case Post-Baseline, To W/in Range or No Change | 1 | 1
  Potassium, Worst Case Post-Baseline, To High | 0 | 0
  Sodium, Worst Case Post-Baseline, To Low | 0 | 0
  Sodium, Worst Case Post-Baseline, To W/in Range or No Change | 1 | 1
  Sodium, Worst Case Post-Baseline, To High | 0 | 0

11. Primary Outcome: Part 2: Cohorts 4: Number of Participants With Worst Case Hematology Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected for analysis of hematology parameters. The ranges for hematology parameters are as follows: Hematocrit[>51 % in male, >45% in female], Haemoglobin[Higher: > 175 grams/Litre (g/L) in male, >150 g/L in female and Low: less than (<) 100 g/L in male, <95 g/L in female], Lymphocytes[<0.97 10^9/L], Neutrophils[<1.5 10^9/L], Platelets[High: > 550 10^9/ L and Low: < 100 10^9/ L], White blood cells[High:>18 10^9/L Low:<2 10^9/L], Red blood cells[Low: <3.0 10^12/L in male, <2.5 10^12/L]. Participants were counted in worst case category that their value changes to (low, within range or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (for example [e.g.], High to High), or whose value became within range, were recorded in "To within Range or No Change" category. Participants were counted twice if participant has values that changed 'To Low' & 'To High', so the percentages may not add to 100%.
Time Frame: Upto Week 9
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 4: Placebo C4 | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1 | 1
Participants
  Erythrocytes, Baseline, Low | 0 | 0
  Erythrocytes, Baseline, W/in Range | 1 | 1
  Erythrocytes, Baseline, High | 0 | 0
  Hematocrit, Baseline, Low | 0 | 0
  Hematocrit, Baseline, W/in Range | 0 | 0
  Hematocrit, Baseline, High | 1 | 1
  Hemoglobin, Baseline, Low | 0 | 0
  Hemoglobin, Baseline, W/in Range | 1 | 1
  Hemoglobin, Baseline, High | 0 | 0
  Leukocytes, Baseline, Low | 0 | 0
  Leukocytes, Baseline, W/in Range | 1 | 1
  Leukocytes, Baseline, High | 0 | 0
  Neutrophils, Baseline, Low | 0 | 0
  Neutrophils, Baseline, W/in Range | 1 | 1
  Neutrophils, Baseline, High | 0 | 0
  Platelets, Baseline, Low | 0 | 0
  Platelets, Baseline, W/in Range | 1 | 1
  Platelets, Baseline, High | 0 | 0

12. Primary Outcome: Part 2: Cohorts 4: Number of Participants With Worst Case Urinalysis Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: Urine samples were collected to assess urine glucose, protein, occult blood and ketones using dipstick method. The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters were recorded as negative, trace, 1+, 2+, 3+ indicating proportional concentrations in the urine sample. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Result for urinalysis parameters were recorded as no change/decreased and any increase.
Time Frame: Upto Week 9
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 4: Placebo C4 | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1 | 1
Participants
  Glucose, No Change/Decreased | 1 | 1
  Ketones, No Change/Decreased | 0 | 1
  Ketones, Increase to TRACE | 1 | 0
  Protein, No Change/Decreased | 1 | 1

13. Primary Outcome: Part 2: Cohorts 4: Number of Participants With Clinically Significant Changes in Hepatobiliary Laboratory Values
Description: Blood samples were collected to evaluate hepatobiliary abnormalities. Number of participants with Bilirubin (BIL), Alkaline phosphatase (ALP), Alanine Aminotransferase (ALT) in combination of these with levels more than the defined hepatobiliary abnormality criteria were presented. Hepatocellular injury is defined as ([ALT/ALT ULN]/[ALP/ALP ULN]) greater than or equal to (>=) 5 and ALT >=3xULN.
Time Frame: Upto Week 9
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 4: Placebo C4 | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1 | 1
Participants
  ALT >=3xULN and BIL >=2xULN | 0 | 0
  ALT >3xULN and BIL >= 2xULN and (ALP <2xULN) | 0 | 0
  ALT >3xULN and INR >1.5: number analyzed (Participants) | 0 | 0
  Hepatocellular injury | 0 | 0
  Hepatocellular injury and BIL >2xULN | 0 | 0
  ALT > 1.5xULN | 0 | 1
  ALT >= 3xULN | 0 | 0
  ALT >= 5xULN | 0 | 0
  ALT >= 8xULN | 0 | 0
  ALT >= 10xULN | 0 | 0
  ALT >= 20xULN | 0 | 0

14. Primary Outcome: Part 2: Cohorts 4: Number of Participants With Clinically Significant Changes in 12-lead ECG Laboratory Values
Description: as for outcome 7
Time Frame: Upto Week 9
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 4: Placebo C4 | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1 | 1
Participants
  Cohort 4 Day -1, Not Clinically Significant | 1 | 0
  Cohort 4 Day -1, Clinically Significant | 0 | 0
  Cohort 4 Day 1, Not Clinically Significant | 1 | 1
  Cohort 4 Day 1, Clinically Significant | 0 | 0
  Cohort 4 Day 2, Not Clinically Significant | 0 | 0
  Cohort 4 Day 2, Clinically Significant | 0 | 0
  Cohort 4 Day 3, Not Clinically Significant | 1 | 1
  Cohort 4 Day 3, Clinically Significant | 0 | 0
  Cohort 4 Day 4, Not Clinically Significant | 0 | 0
  Cohort 4 Day 4, Clinically Significant | 0 | 0
  Cohort 4 Day 5, Not Clinically Significant | 0 | 0
  Cohort 4 Day 5, Clinically Significant | 0 | 0
  Cohort 4 Day 6, Not Clinically Significant | 0 | 0
  Cohort 4 Day 6, Clinically Significant | 0 | 0
  Cohort 4 Day 7, Not Clinically Significant | 0 | 0
  Cohort 4 Day 7, Clinically Significant | 0 | 0
  Cohort 4 Day 8, Not Clinically Significant | 0 | 0
  Cohort 4 Day 8, Clinically Significant | 0 | 0
  Cohort 4 Day 9, Not Clinically Significant | 0 | 0
  Cohort 4 Day 9, Clinically Significant | 0 | 0
  Cohort 4 Day 10, Not Clinically Significant | 0 | 0
  Cohort 4 Day 10, Clinically Significant | 0 | 0
  Cohort 4 Day 11, Not Clinically Significant | 0 | 0
  Cohort 4 Day 11, Clinically Significant | 0 | 0
  Cohort 4 Day 12, Not Clinically Significant | 0 | 0
  Cohort 4 Day 12, Clinically Significant | 0 | 0
  Cohort 4 Day 13, Not Clinically Significant | 1 | 0
  Cohort 4 Day 13, Clinically Significant | 0 | 0
  Cohort 4 Day 14, Not Clinically Significant | 1 | 1
  Cohort 4 Day 14, Clinically Significant | 0 | 0
  Cohort 4 Day 15, Not Clinically Significant | 0 | 0
  Cohort 4 Day 15, Clinically Significant | 0 | 0
  Cohort 4 Day 16, Not Clinically Significant | 0 | 0
  Cohort 4 Day 16, Clinically Significant | 0 | 0
  Cohort 4 Day 17, Not Clinically Significant | 0 | 0
  Cohort 4 Day 17, Clinically Significant | 0 | 0
  Cohort 4 Day 18, Not Clinically Significant | 0 | 0
  Cohort 4 Day 18, Clinically Significant | 0 | 0
  Cohort 4 Day 19, Not Clinically Significant | 0 | 0
  Cohort 4 Day 19, Clinically Significant | 0 | 0
  Worst Case Post Baseline, Not Clinically Significant | 1 | 1
  Worst Case Post Baseline, Clinically Significant | 0 | 0

15. Primary Outcome: Part 2: Cohorts 4: Number of Participants With Worst Case Vital Signs Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: as for outcome 8
Time Frame: Upto Week 9
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 4: Placebo C4 | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1 | 1
Participants
  DBP, Period 1 Worst Case Post Baseline, To Low | 0 | 0
  DBP, Period 1 Worst Case Post Baseline, To w/in Range or No Change | 1 | 1
  DBP, Period 1 Worst Case Post Baseline, To High | 0 | 0
  PR, Period 1 Worst Case Post Baseline, To Low | 0 | 0
  PR, Period 1 Worst Case Post Baseline, To w/in Range or No Change | 1 | 1
  PR, Period 1 Worst Case Post Baseline, To High | 0 | 0
  Systolic Blood Pressure, Period 1 Worst Case Post Baseline, To Low | 0 | 0
  Systolic Blood Pressure, Period 1 Worst Case Post Baseline, To w/in Range or No Change | 1 | 1
  Systolic Blood Pressure, Period 1 Worst Case Post Baseline, To High | 0 | 0
  RR, Period 1 Worst Case Post Baseline, To Low | 0 | 0
  RR, Period 1 Worst Case Post Baseline, To w/in Range or No Change | 1 | 1
  RR, Period 1 Worst Case Post Baseline, To High | 0 | 0
  Temperature, Period 1 Worst Case Post Baseline, To Low | 0 | 0
  Temperature, Period 1 Worst Case Post Baseline, To w/in Range or No Change | 1 | 1
  Temperature, Period 1 Worst Case Post Baseline, To High | 0 | 0

16. Primary Outcome: Part 2: Cohorts 4: Number of Participants With Clinically Significant Changes in Echocardiogram
Description: Echocardiography was performed at screening and Part 2 of the study using sound waves.
Time Frame: Upto Week 9
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 4: Placebo C4 | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

17. Primary Outcome: Part 2: Cohorts 4: Number of Participants With Clinically Significant Changes in Continuous Telemetry
Description: as for outcome 9
Time Frame: Upto Day 14
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 4: Placebo C4 | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1 | 1
Participants
  Cohort 4 Day 2, Not Clinically Significant | 1 | 0
  Cohort 4 Day 2, Clinically Significant | 0 | 0
  Cohort 4 Day 3, Not Clinically Significant | 1 | 0
  Cohort 4 Day 3, Clinically Significant | 0 | 0
  Cohort 4 Day 4, Not Clinically Significant | 1 | 0
  Cohort 4 Day 4, Clinically Significant | 0 | 0
  Cohort 4 Day 5, Not Clinically Significant | 1 | 0
  Cohort 4 Day 5, Clinically Significant | 0 | 0
  Cohort 4 Day 6, Not Clinically Significant | 1 | 0
  Cohort 4 Day 6, Clinically Significant | 0 | 0
  Cohort 4 Day 7, Not Clinically Significant | 1 | 0
  Cohort 4 Day 7, Clinically Significant | 0 | 0
  Cohort 4 Day 8, Not Clinically Significant | 1 | 0
  Cohort 4 Day 8, Clinically Significant | 0 | 0
  Cohort 4 Day 9, Not Clinically Significant | 1 | 0
  Cohort 4 Day 9, Clinically Significant | 0 | 0
  Cohort 4 Day 10, Not Clinically Significant | 1 | 0
  Cohort 4 Day 10, Clinically Significant | 0 | 0
  Cohort 4 Day 11, Not Clinically Significant | 1 | 0
  Cohort 4 Day 11, Clinically Significant | 0 | 0
  Cohort 4 Day 12, Not Clinically Significant | 1 | 0
  Cohort 4 Day 12, Clinically Significant | 0 | 0
  Cohort 4 Day 13, Not Clinically Significant | 1 | 0
  Cohort 4 Day 13, Clinically Significant | 0 | 0
  Cohort 4 Day 15, Not Clinically Significant | 1 | 0
  Cohort 4 Day 15, Clinically Significant | 0 | 0
  Worst Case Post Baseline, Not Clinically Significant | 1 | 0
  Worst Case Post Baseline, Clinically Significant | 0 | 0

18. Primary Outcome: Part 1: Area Under the Plasma Concentration Curve From Time Zero to Last Time of Quantifiable Concentration (AUC[0-t]) of GSK3884464 Following Single Dose Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of AUC[0-t].
Time Frame: Day 1 pre-dose,15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, and 120 hours post-dose
Population: The analysis was performed on the Pharmacokinetic (PK) Set that includes all participants in the Safety population who had at least one non-missing PK assessment (Non-quantifiable [NQ] values were considered as valid PK assessment). This population was based on the treatment the participant actually received. Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Picograms Per Milliliter (h*pg/mL)
Arm/Group | Part 1 Cohort 1: GSK3884464 1 mg | Part 1 Cohort 1: GSK3884464 3 mg | Part 1 Cohort 1: GSK3884464 9 mg | Part 1 Cohort 2: GSK3884464 30 mg | Part 1 Cohort 2: GSK3884464 110 mg | Part 1 Cohort 3: GSK3884464 70 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 1
Hour*Picograms Per Milliliter (h*pg/mL) | 1031.06 (35.88) | 3104.28 (27.33) | 8510.99 (30.70) | 23966.53 (24.35) | 76886.06 (11.20) | 99220.48 (NA) — NA indicates geometric coefficient of variation could not be calculated for single participant.

19. Primary Outcome: Part 1: AUC From Time Zero to Infinity (AUC[0-inf]) of GSK3884464 Following Single Dose Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of AUC[0-t].
Time Frame: Day 1 pre-dose,15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, and 120 hours post-dose
Population: The analysis was performed on the PK Set that includes all participants in the Safety population who had at least one non-missing PK assessment (Non-quantifiable [NQ] values were considered as valid PK assessment). This population was based on the treatment the participant actually received. Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Picograms Per Milliliter (h*pg/mL)
Arm/Group | Part 1 Cohort 1: GSK3884464 1 mg | Part 1 Cohort 1: GSK3884464 3 mg | Part 1 Cohort 1: GSK3884464 9 mg | Part 1 Cohort 2: GSK3884464 30 mg | Part 1 Cohort 2: GSK3884464 110 mg | Part 1 Cohort 3: GSK3884464 70 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 1
Hour*Picograms Per Milliliter (h*pg/mL) | 1177.89 (39.36) | 3422.89 (32.86) | 9632.76 (36.64) | 27096.66 (28.90) | 81971.94 (11.22) | 101162.62 (NA) — NA indicates geometric coefficient of variation could not be calculated for single participant.

20. Primary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of GSK3884464 Following Single Dose Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of Cmax.
Time Frame: Day 1 pre-dose,15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, and 120 hours post-dose
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms Per Milliliter (ng/mL)
Arm/Group | Part 1 Cohort 1: GSK3884464 1 mg | Part 1 Cohort 1: GSK3884464 3 mg | Part 1 Cohort 1: GSK3884464 9 mg | Part 1 Cohort 2: GSK3884464 30 mg | Part 1 Cohort 2: GSK3884464 110 mg | Part 1 Cohort 3: GSK3884464 70 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 3 | 1
Nanograms Per Milliliter (ng/mL) | 70.69 (17.52) | 211.56 (23.51) | 551.75 (23.60) | 1892.92 (36.46) | 5093.44 (22.38) | 6650.00 (NA) — NA indicates geometric coefficient of variation could not be calculated for single participant.

21. Primary Outcome: Part 1: Time to Maximum Observed Plasma Drug Concentration (Tmax) of GSK3884464 Following Single Dose Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of Tmax.
Time Frame: Day 1 pre-dose,15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, and 120 hours post-dose
Population: as for outcome 19
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Part 1 Cohort 1: GSK3884464 1 mg | Part 1 Cohort 1: GSK3884464 3 mg | Part 1 Cohort 1: GSK3884464 9 mg | Part 1 Cohort 2: GSK3884464 30 mg | Part 1 Cohort 2: GSK3884464 110 mg | Part 1 Cohort 3: GSK3884464 70 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 3 | 1
Hour (h) | 0.51 [0.49 to 1.00] | 1.0 [0.51 to 1.01] | 1.01 [0.50 to 1.50] | 1.00 [0.50 to 4.00] | 1.51 [1.02 to 1.51] | 2.00 [2.00 to 2.00]

22. Primary Outcome: Part 1: Terminal Half-life (T1/2) of GSK3884464 Following Single Dose Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of T1/2.
Time Frame: Day 1 pre-dose,15, 30 minutes, 1, 1.5, 2, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, and 120 hours post-dose
Population: as for outcome 19
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Part 1 Cohort 1: GSK3884464 1 mg | Part 1 Cohort 1: GSK3884464 3 mg | Part 1 Cohort 1: GSK3884464 9 mg | Part 1 Cohort 2: GSK3884464 30 mg | Part 1 Cohort 2: GSK3884464 110 mg | Part 1 Cohort 3: GSK3884464 70 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 3 | 1
Hour (h) | 38.87 [28.78 to 76.10] | 32.39 [21.02 to 71.75] | 37.58 [26.90 to 76.11] | 31.845 [23.31 to 77.52] | 31.49 [21.29 to 39.50] | 21.50 [21.50 to 21.50]

23. Primary Outcome: Part 2: Cohorts 4: AUC Over the Dosing Interval (AUC[Tau]) of GSK3884464 Following Repeat Dose Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of AUC [tau] for repeat dose administration. NA indicates geometric coefficient of variation could not be calculated for single participant.
Time Frame: Day 1: pre-dose, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24 hours post-dose; Day 4 and Day 11: pre-dose; Day 7: pre-dose, 6 and 12 hours post-dose; Day 14: pre-dose, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96 and 120 hours post-dose
Population: The analysis was performed on the PK Set that includes all participants in the Safety population who had at least one non-missing PK assessment (Non-quantifiable [NQ] values were considered as valid PK assessment). This population was based on the treatment the participant actually received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Picograms Per Milliliter (h*pg/mL)
Arm/Group | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1
Hour*Picograms Per Milliliter (h*pg/mL) | 11902.86 (NA) — NA indicates geometric coefficient of variation could not be calculated for single participant

24. Primary Outcome: Part 2: Cohorts 4: Cmax of GSK3884464 Following Repeat Dose Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of Cmax for repeat dose administration. NA indicates geometric coefficient of variation could not be calculated for single participant.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms Per Milliliter (ng/mL)
Arm/Group | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1
Nanograms Per Milliliter (ng/mL)
  Cohort 4 Day 1 | 754.00 (NA) — NA indicates geometric coefficient of variation could not be calculated for single participant
  Cohort 4 Day 14 | 1120.00 (NA) — NA indicates geometric coefficient of variation could not be calculated for single participant

25. Primary Outcome: Part 2: Cohorts 4: Trough Plasma Concentration (Ctau) of GSK3884464 Following Repeat Dose Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of Ctau for repeat dose administration. NA indicates geometric coefficient of variation could not be calculated for single participant.
Time Frame: as for outcome 23
Population: The analysis was performed on the PK Set that includes all participants in the Safety population who had at least one non-missing PK assessment (NQ values were considered as valid PK assessment). This population was based on the treatment the participant actually received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms Per Milliliter (ng/mL)
Arm/Group | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1
Nanograms Per Milliliter (ng/mL)
  Cohort 4 Day 1 | 246.00 (NA) — NA indicates geometric coefficient of variation could not be calculated for single participant.
  Cohort 4 Day 14 | 415.99 (NA) — NA indicates geometric coefficient of variation could not be calculated for single participant.

26. Primary Outcome: Part 2: Cohorts 4: Tmax of GSK3884464 Following Repeat Dose Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of Tmax for repeat dose administration. NA indicates full range could not be calculated for single participant.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1
Hour (h)
  Cohort 4 Day 1 | 0.57 [NA to NA] — NA indicates full range could not be calculated for single participant.
  Cohort 4 Day 14 | 0.57 [NA to NA] — NA indicates full range could not be calculated for single participant.

27. Primary Outcome: Part 2: Cohorts 4: T1/2 of GSK3884464 Following Repeat Dose Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of T1/2 for repeat dose administration. NA indicates full range could not be calculated for single participant.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1
Hour (h)
  Cohort 4 Day 1 | 70.59 [NA to NA] — NA indicates full range could not be calculated for single participant.
  Cohort 4 Day 14 | 45.05 [NA to NA] — NA indicates full range could not be calculated for single participant.

28. Primary Outcome: Part 2: Cohorts 4: Accumulation Ratio Based on AUC(Tau) (RAUC) of GSK3884464 Following Repeat Dose Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of RAUC for repeat dose administration. NA indicates geometric coefficient of variation could not be calculated for single participant.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1
Ratio | 1.77 (NA) — NA indicates geometric coefficient of variation could not be calculated for single participant

29. Primary Outcome: Part 2: Cohorts 4: Accumulation Ratio Based on Cmax (RCmax) of GSK3884464 Following Repeat Dose Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of RCmax for repeat dose administration. NA indicates geometric coefficient of variation could not be calculated for single participant.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1
Ratio | 1.49 (NA) — NA indicates geometric coefficient of variation could not be calculated for single participant

30. Primary Outcome: Part 2: Cohorts 4: Accumulation Ratio Based on Ctau (RCtau) of GSK3884464 Following Repeat Dose Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of RCtau for repeat dose administration. NA indicates geometric coefficient of variation could not be calculated for single participant.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1
Ratio | 1.68 (NA) — NA indicates geometric coefficient of variation could not be calculated for single participant.

31. Secondary Outcome: Part 1: Change From Baseline in NAD(P)H Dehydrogenase Quinone 1 (NQO1) Messenger Ribonucleic Acid (mRNA) in Whole Blood Post Treatment With GSK3884464
Description: Blood samples were collected at indicated time points for pharmacodynamic analysis of NQO1 mRNA.
Time Frame: Day1: pre-dose,30 minutes,1,1.5,2,3,4,6, 8,12,18,24 hours post-dose
Population: The analysis was performed on the Pharmacodynamic (PD) Set that includes all participants in the Safety population with baseline and at least one post baseline PD measure (e.g., NQO1 mRNA). Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Fold Change
Arm/Group | Part 1 Cohort 1: Placebo C1 | Part 1 Cohort 1: GSK3884464 1 mg | Part 1 Cohort 1: GSK3884464 3 mg | Part 1 Cohort 1: GSK3884464 9 mg | Part 1 Cohort 2: Placebo C2 | Part 1 Cohort 2: GSK3884464 30 mg | Part 1 Cohort 2: GSK3884464 110 mg | Part 1 Cohort 3: Placebo C3 | Part 1 Cohort 3: GSK3884464 70 mg
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 5 | 6 | 3 | 1 | 1
Fold Change | 1.19 (0.17) | 1.17 (0.11) | 1.13 (0.10) | 1.31 (0.29) | 1.16 (0.20) | 2.79 (0.69) | 7.66 (1.52) | 0.96 (NA) — NA indicates standard deviation could not be calculated for single participant. | 8.5830 (NA) — NA indicates standard deviation could not be calculated for single participant.

32. Secondary Outcome: Part 2: Cohorts 4: Change From Baseline in NQO1 mRNA in Whole Blood Post Treatment With GSK3884464
Description: Blood samples were collected at indicated time points for pharmacodynamic analysis of NQO1 mRNA for repeat dose administration. NA indicates standard deviation could not be calculated for single participant.
Time Frame: as for outcome 23
Population: The analysis was performed on the PD Set that includes all participants in the Safety population with baseline and at least one post baseline PD measure (e.g., NQO1 mRNA).
Measure: Mean (Standard Deviation); unit: Fold Change
Arm/Group | Part 2 Cohort 4: Placebo C4 | Part 2 Cohort 4: GSK3884464 15 mg
Number analyzed (Participants) | 1 | 1
Fold Change
  Cohort 4 Day 1 | 1.035 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | 1.684 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.
  Cohort 4 Day 7 | 1.095 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | 2.560 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.
  Cohort 4 Day 14 | 1.029 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | 2.405 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were collected up to Day 17 for Cohort 1, 2 and 3 of Part 1, up to Day 29 for Cohort 4 of Part 2.
Description: Safety Set comprised of all randomized participants who received at least 1 dose of study intervention.
Arm/Group | Part 1 Cohort 1: Placebo C1 | Part 1 Cohort 1: GSK3884464 1 mg | Part 1 Cohort 1: GSK3884464 3 mg | Part 1 Cohort 1: GSK3884464 9 mg | Part 1 Cohort 2: Placebo C2 | Part 1 Cohort 2: GSK3884464 30 mg | Part 1 Cohort 2: GSK3884464 110 mg | Part 1 Cohort 3: Placebo C3 | Part 1 Cohort 3: GSK3884464 70 mg | Part 2 Cohort 4: Placebo C4 | Part 2 Cohort 4: GSK3884464 15 mg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/3 | 0/1 | 0/1 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6 | 1/5 | 0/6 | 0/3 | 0/1 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 2/9 | 1/6 | 0/6 | 3/6 | 3/5 | 1/6 | 3/3 | 1/1 | 1/1 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Cohort 1: Placebo C1 (N=9) | Part 1 Cohort 1: GSK3884464 1 mg (N=6) | Part 1 Cohort 1: GSK3884464 3 mg (N=6) | Part 1 Cohort 1: GSK3884464 9 mg (N=6) | Part 1 Cohort 2: Placebo C2 (N=5) | Part 1 Cohort 2: GSK3884464 30 mg (N=6) | Part 1 Cohort 2: GSK3884464 110 mg (N=3) | Part 1 Cohort 3: Placebo C3 (N=1) | Part 1 Cohort 3: GSK3884464 70 mg (N=1) | Part 2 Cohort 4: Placebo C4 (N=1) | Part 2 Cohort 4: GSK3884464 15 mg (N=1)
Albuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Cohort 1: Placebo C1 (N=9) | Part 1 Cohort 1: GSK3884464 1 mg (N=6) | Part 1 Cohort 1: GSK3884464 3 mg (N=6) | Part 1 Cohort 1: GSK3884464 9 mg (N=6) | Part 1 Cohort 2: Placebo C2 (N=5) | Part 1 Cohort 2: GSK3884464 30 mg (N=6) | Part 1 Cohort 2: GSK3884464 110 mg (N=3) | Part 1 Cohort 3: Placebo C3 (N=1) | Part 1 Cohort 3: GSK3884464 70 mg (N=1) | Part 2 Cohort 4: Placebo C4 (N=1) | Part 2 Cohort 4: GSK3884464 15 mg (N=1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT05044325/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT05044325/SAP_001.pdf